CLINICAL TRIAL: NCT00269542
Title: Impact of Zinc Supplementation on Mortality and Hospitalizations in Children Aged 1 Months to 23 Months
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Society for Applied Studies (Other)
Collaborators: World Health Organization (Other); All India Institute of Medical Sciences (Other)
Responsible Party: Dr. MK Bhan, All India Institute of Medical Sciences
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 00002; C6-181-429
Record Dates: First submitted 2005-12-22; First posted 2005-12-23 (Estimated); Last update posted 2008-07-01 (Estimated); Status verified 2008-06

CONDITIONS: Morbidity; Mortality; Diarrhea; Pneumonia
Keywords: zinc supplementation; hospitalisations; children; mortality; iron folic acid
MeSH Terms: conditions — Diarrhea; Pneumonia | interventions — Zinc

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Zinc and iron folic acid - Intervention
- 2 (Placebo Comparator)
  Interventions: Drug: Iron Folic Acid alone - Placebo

INTERVENTIONS:
Drug: Zinc and iron folic acid - Intervention — The intervention group tablet contained 10 mg of elemental zinc, 12.5 mg of iron and 50 micrograms of folic acid.
  Arms: 1
Drug: Iron Folic Acid alone - Placebo — The control group tablets were similar in composition, appearance and taste except it contained placebo for zinc.
  Arms: 2

SUMMARY:
Children, aged 1 months to 23 months, in the intervention households received zinc, iron and folic acid and those in the control households were administered iron and folic acid (IFA) alone for a period of one year. The primary outcomes were hospitalizations and deaths during this period.

DETAILED DESCRIPTION:
Objective: Studies in developing countries show substantial reduction in diarrhoea and respiratory morbidity in young children receiving zinc supplementation. The impact of daily zinc supplementation coadministered with iron folic acid in young children on all cause hospitalisation and mortality in comparison with iron folic acid alone, was evaluated to help shape public policy.

Design: Randomised double blind trial

Setting: Low to middle socio-economic urban neighbourhoods of north and north-west Delhi in India

Participants: 94359 subjects aged 1 month to 23 months

Interventions: The subjects were administered dispersible tablets containing one recommended daily allowance of zinc and iron folic acid or iron folic acid alone, daily for 12 months after enrolment.

Main outcome measures: Hospitalisations were captured through passive surveillance of eight hospitals by trained study physicians. Deaths were ascertained through bimonthly visits to households.

Results: A third of the total children had low zinc levels (<60 mg/dL) and one fourth had iron deficiency (haematocrit <33%) at baseline. The proportion zinc deficient was significantly lower post 12 months supplementation, in the zinc and iron folic acid group (difference in proportions -10%; 95% confidence interval -15.6% to -4.4%, p 0.0005). Only 7.7% in the zinc and iron folic acid and 7.3% in the iron folic acid group had low haematocrit. Zinc and iron folic acid supplementation had no impact on hospitalisations, overall and cause-specific. The overall death rates were similar in the two groups.

Conclusions: The lack of mortality impact may be real or the findings could have resulted from the use of lower daily zinc dosing than in morbidity prevention trials or an interaction between zinc and iron whereby adding iron, may have adversely affected potential effects of zinc on immune function and morbidity. Future research should address iron and zinc interaction effects on important functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 1 months to 23 months
* Either sex
* Resident of study area

Exclusion Criteria:

* Likely to leave the area during the study period
* Non consent
* Temporary exclusion criteria Illness requiring hospitalization Visible severe wasting. Visibly wasted children will be referred to a hospital for treatment. They will be eligible for enrollment only after effective rehabilitation.

Ages: 1 Month to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 94359 (Actual)
Dates: Start 2002-02; Primary Completion 2003-03 (Actual); Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
- to determine the impact of daily oral supplementation of zinc (5 mg per day to infants aged less than 6 months and 10 mg per day to older children) and iron folic acid to children aged 1-23 months for a period of upto 12 months on all-cause mortality, | 3 monthly home visits
- to determine the impact of daily oral supplementation of zinc and iron folic acid to children 1-23 months for a period of upto 12 months on overall and diarrhea and pneumonia specific hospital admissions. | 3 monthly home visits

SECONDARY OUTCOMES:
- the proportion of stunted or underweight children at end study | Baseline and end study after 12 months
- the proportion of zinc deficient (plasma zinc <60 mg/dl) children at end study | Baseline and end study after 12 months
- the mean plasma copper and superoxide dismutase at end study | Baseline and end study after 12 months
- the mean plasma ferritin and transferrin activity at end study | Baseline and end study after 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Maharaj K Bhan, MD, Principal Investigator — Professor, Department of Pediatrics, All India Institute of Medical Sciences; Nita Bhandari, PhD, Principal Investigator — Society for Applied Studies, New Delhi

REFERENCES:
- [Background] Bhandari N, Taneja S, Mazumder S, Bahl R, Fontaine O, Bhan MK; Zinc Study Group. Adding zinc to supplemental iron and folic acid does not affect mortality and severe morbidity in young children. J Nutr. 2007 Jan;137(1):112-7. doi: 10.1093/jn/137.1.112. PMID 17182810